CLINICAL TRIAL: NCT04086797
Title: Double-blind, Randomised, Placebo-controlled Study to Evaluate the Efficacy and Safety of IQP-AE-103 in Overweight and Moderately Obese Subjects
Brief Title: DBRPC Study to Evaluate the Efficacy and Safety of IQP-AE-103 in Overweight and Moderately Obese Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Perrigo CSCI (Industry)
Collaborators: Analyze & Realize (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PERI/020918
Record Dates: First submitted 2019-09-10; First posted 2019-09-12 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Overweight; Obesity
Keywords: IQP-AE-103; overweight treatment; obesity treatment
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IQP-AE-103 (Experimental): 2 capsules after 3 main meals per day (total 1980 mg)
  Interventions: Dietary Supplement: IQP-AE-103
- Placebo (Placebo Comparator): 2 capsules after 3 main meals per day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: IQP-AE-103 — 1980 mg
  Arms: IQP-AE-103
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The main study objective is to evaluate the efficacy of IQP-AE-103 in reducing body weight in overweight and moderately obese subjects, in the context of an energy restricted diet. Further objectives are to evaluate the beneficial potential of IQP-AE-103 on waist circumference, blood pressure and blood glucose and lipid levels, quality of life, as well as its safety and tolerability

DETAILED DESCRIPTION:
Overweight and obesity are defined as abnormal or excessive fat accumulation that may impair health. Obesity is a substantial public health problem throughout the world, with the prevalence increasing rapidly in numerous developing and developed nations. In 2014, about 13% of the world's adult populations were obese and 39% were overweight. The worldwide prevalence of obesity has more than doubled in over 30 years (WHO, 2016). Obesity and overweight pose major risks for serious diseases, such as dyslipidemia, type 2 diabetes, hypertension, coronary heart disease and stroke (Haslam & James 2005) and average life expectancy is reduced in obese people (Fontaine et al. 2003). Dietary fat plays a major role in the development of overeating and obesity (Bray et al. 2004); thus fat uptake should be a main target to reduce energy intake and achieve a loss of body weight (Svendsen & Tonstad, 2011). It has been shown that nutrients such as protein and fibre reduce lipid absorption (e.g. Chong et al., 2014; Hosomi et al., 2010; Tsujita et al., 2007). The main components of the IQP-AE-103 are okra (Abelmoschus esculentus (L.) Moench) pod powder and inulin. Okra pod powder contains a combination of dietary fibre and protein, which may have an important role in fat binding (Kumar et al., 2013). Dehydrated powder derived from okra pod has further been shown to have substantial swelling capabilities when added to water (Bakre & Jaiyeaob, 2009), which can potentially provide satiety effects. Inulin is a fermentable fructan, derived from plants such as asparagus, garlic, leak, onion etc.

and serves as an important source of soluble dietary fibre (Jaundzeikare and Beitane, 2014), to further enhance the effect of fat binding. The efficacy of IQP-AE-103 in body weight reduction during intake of 12 weeks has been shown recently in a clinical trial with 108 overweight and moderately obese subjects (Uebelhack et al., 2019). The present study aims at a broader evaluation of the beneficial effects of IQP-AE-103 for use in weight management, including its impact on waist circumference, blood pressure and blood glucose and lipid levels as well as quality of life, in overweight and moderately obese subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women from 18 to 70 years old
2. Body mass index (BMI) 25 kg/m2 - 34.9 kg/m2
3. Having at least one of the following traits:

   * waist circumference ≥ 94 cm in men and ≥ 80 cm in women
   * triglyceride levels ≥ 150 mg/dL (1.7 mmol/L)
   * high-density lipoprotein cholesterol (HDL-C) levels: ≤ 40 mg/dL (1.0 mmol/L) in men and ≤ 50 mg/dL (1.3 mmol/L) in women
   * blood pressure (BP), average value of the last two values of the triplicate measurement: systolic BP ≥ 130 mmHg, diastolic BP ≥ 85 mmHg
   * fasting blood glucose ≥ 100 mg/dL
4. Desire to lose weight
5. Readiness and ability to complete the study, according to investigator's judgement following the screening interview
6. Accustomed to regular daily consumption of 3 main meals (breakfast, lunch, dinner)
7. Consistent and stable body weight in the last 3 months prior to V1 (less than 5% self-reported change)
8. Subject's agreement to comply with study procedures, in particular:

   * to adhere to diet recommendation during the study
   * to take IP as recommended
   * to avoid the use of other weight loss and/or management products and/or programs during the study
   * to keep the habitual level of physical activity
   * to complete the subject diary and study questionnaires
9. Women of childbearing potential:

   * commitment to use contraception methods
   * negative pregnancy testing (beta human chorionic gonadotropin test in urine) at V1
10. Readiness not to participate in another clinical study during this study Participation is based upon written informed consent by the participant following written and oral information by the investigator regarding nature, purpose, consequences and possible risks of the clinical study.

Exclusion Criteria:

1. Known allergy or hypersensitivity to the components of the investigational product or source plants
2. Pathological electrocardiogram (ECG) at V1
3. History and/or presence of clinically significant condition/ disorder, which per investigator's judgement could interfere with the results of the study or the safety of the subject, e.g.:

   * untreated or unstable thyroid gland disorder
   * hypertension (regular systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg)
   * acute or chronic gastrointestinal (GI) disease or digestion/ absorption disorders (e.g. inflammatory bowel disease, coeliac disease, pancreatitis etc.)
   * diabetes mellitus
   * any other relevant serious organ or systemic diseases
4. Significant surgery within the last 6 months prior to V1 or planned within the study period:

   * GI surgery
   * liposuction
5. History of eating disorders like bulimia, anorexia nervosa, binge-eating within the last 12 months prior to V1
6. Deviation of safety laboratory parameter(s) at V1 (excluding those stated in the inclusion criteria) that is:

   * clinically significant or
   * >2x upper limit of normal, unless the deviation is justified by a previously known not clinically relevant condition (e.g. Gilbert's syndrome)
7. Any electronic medical implant
8. Regular medication and/or supplementation and/or treatment within the last 3 months prior to V1 and during the study:

   * that could influence body weight (e.g. systemic corticosteroids)
   * that could influence gastrointestinal functions (e.g. laxatives, opioids, anticholinergics etc.) as per investigator judgement
   * for weight management (e.g. fat binder, carbohydrate/ starch blocker, fat burner, satiety products, acupuncture etc.)
   * that could influence lipid levels, blood pressure and/or glycemic control
9. Self-reported smoking cessation within 6 months prior to V1 and/or during the study (regular smoking during the study at the same level as prior to the study is allowed)
10. Women of child-bearing potential: pregnancy or nursing
11. History of or current abuse of drugs, alcohol or medication
12. Participation in another study during the last 30 days prior to V1
13. Any other reason for exclusion as per investigator's judgment, e.g. insufficient compliance with study procedures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2021-04-08 (Actual)

PRIMARY OUTCOMES:
Difference in body weight | 24 weeks
  Difference in body weight (kg) change after 24 weeks of IP intake, in comparison to baseline

SECONDARY OUTCOMES:
Difference in BMI | 24 weeks
  Difference in BMI change after 24 weeks of IP intake, in comparison to baseline

OTHER OUTCOMES:
Difference in change in waist circumference after 24 weeks weeks of IP intake, in comparison to baseline | 24 weeks
  weeks of IP intake, in comparison to baseline
Difference in body weight (%) change after 24 weeks of IP intake, in comparison to baseline | 24 weeks
  Difference in body weight (%) change after 24 weeks
Difference in body weight (kg) change after 16 weeks of IP intake, in comparison to baseline | 16 weeks
  Difference in body weight (kg) change after 16 weeks
Difference in body weight (%) change after 16 weeks of IP intake, in comparison to baseline | 16 weeks
  Difference in body weight (%) change after 16 weeks
Difference in BMI change after 16 weeks of IP intake, in comparison to baseline | 16 weeks
  Difference in BMI change after 16 weeks of IP intake,
Difference in body fat mass (kg) change assessed per BIA after 24 weeks of IP intake, in comparison to baseline | 24 weeks
  Difference in body fat mass (kg) change assessed per BIA after 24 weeks of IP intake, in comparison to baseline
Difference in change in quality of life parameters assessed per IWQOL-LITE after 24 weeks of IP intake, in comparison to baseline | 24 weeks
  Difference in change in quality of life parameters assessed per IWQOL-LITE after 24 weeks of IP intake, in comparison to baseline
Difference in body fat mass (kg) change assessed per BIA after 16 weeks of IP intake, in comparison to baseline | 16 weeks
  Difference in body fat mass (kg) change assessed per BIA after 16 weeks of IP intake, in comparison to baseline
Difference in change in quality of life parameters assessed per IWQOL-LITE after 16 weeks of IP intake, in comparison to baseline | 16 weeks
  Difference in change in quality of life parameters assessed per IWQOL-LITE after 16 weeks of IP intake, in comparison to baseline
Difference in change in systolic blood pressure after 24 weeks of IP intake, in comparison to baseline | 24 weeks
  Difference in change in systolic blood pressure after 24 weeks of IP intake, in comparison to baseline
Difference in change in diastolic blood pressure after 24 weeks of IP intake, in comparison to baseline | 24 weeks
  Difference in change in diastolic blood pressure after 24 weeks of IP intake, in comparison to baseline
Difference in global evaluation of efficacy by subject and investigator at study end | 24 weeks
  Difference in global evaluation of efficacy by subject and investigator at study end
Difference in evaluation of success with respect to the original goal/motivation of the subject to participate at study end | 24 weeks
  Difference in evaluation of success with respect to the original goal/motivation of the subject to participate at study end
Difference in change in waist circumference after 16 weeks of IP intake, in comparison to baseline | 16 weeks
  Difference in change in waist circumference after 16 weeks of IP intake, in comparison to baseline
Difference in change in systolic blood pressure after 16 weeks of IP intake, in comparison to baseline | 16 weeks
  Difference in change in systolic blood pressure after 16 weeks of IP intake, in comparison to baseline
Difference in change in diastolic blood pressure after 16 weeks of IP intake, in comparison to baseline | 16 weeks
  Difference in change in diastolic blood pressure after 16 weeks of IP intake, in comparison to baseline
Difference in change in TG after 24 weeks of IP intake, in comparison to baseline | 24 weeks
  Difference in change in TG after 24 weeks of IP intake, in comparison to baseline
Difference in change in HDL-C after 24 weeks of IP intake, in comparison to baseline | 24 weeks
  Difference in change in HDL-C after 24 weeks of IP intake, in comparison to baseline
Difference in change in LDL-C after 24 weeks of IP intake, in comparison to baseline | 24 weeks
  Difference in change in LDL-C after 24 weeks of IP intake, in comparison to baseline
Difference in change in TC after 24 weeks of IP intake, in comparison to baseline | 24 weeks
  Difference in change in TC after 24 weeks of IP intake, in comparison to baseline
Difference in change in fasting blood glucose after 24 weeks of IP intake, in comparison to baseline | 24 weeks
  Difference in change in fasting blood glucose after 24 weeks of IP intake, in comparison to baseline
Difference in body weight (kg) change after 8 weeks of IP intake, in comparison to baseline | 8 weeks
  Difference in body weight (kg) change after 8 weeks of IP intake, in comparison to baseline
Difference in body weight (%) change after 8 weeks of IP intake, in comparison to baseline | 8 weeks
  Difference in body weight (%) change after 8 weeks of IP intake, in comparison to baseline
Difference in BMI change after 8 weeks of IP intake, in comparison to baseline | 8 weeks
  Difference in BMI change after 8 weeks of IP intake, in comparison to baseline
Difference in body fat mass (kg) change assessed per BIA after 8 weeks of IP intake, in comparison to baseline | 8 weeks
  Difference in body fat mass (kg) change assessed per BIA after 8 weeks of IP intake, in comparison to baseline
Difference in change in quality of life parameters assessed per IWQOL-LITE after 8 weeks of IP intake, in comparison to baseline | 24 weeks
  Difference in change in quality of life parameters assessed per IWQOL-LITE after 8 weeks of IP intake, in comparison to baseline
Difference in change in waist circumference after 8 weeks of IP intake, in comparison to baseline | 8 weeks
  Difference in change in waist circumference after 8 weeks of IP intake, in comparison to baseline
Difference in body weight (kg) change after 4 weeks of IP intake, in comparison to baseline | 4 weeks
  Difference in body weight (kg) change after 4 weeks of IP intake, in comparison to baseline
Difference in body weight (%) change after 4 weeks of IP intake, in comparison to baseline | 4 weeks
  Difference in body weight (%) change after 4 weeks of IP intake, in comparison to baseline
Difference in BMI change after 4 weeks of IP intake, in comparison to baseline | 4 weeks
  Difference in BMI change after 4 weeks of IP intake, in comparison to baseline
Difference in change in systolic blood pressure after 8 weeks of IP intake, in comparison to baseline | 8 weeks
  Difference in change in systolic blood pressure after 8 weeks of IP intake, in comparison to baseline
Difference in change in diastolic blood pressure after 8 weeks of IP intake, in comparison to baseline | 8 weeks
  Difference in change in diastolic blood pressure after 8 weeks of IP intake, in comparison to baseline
Difference in change in TG after 16 weeks of IP intake, in comparison to baseline | 16 weeks
  Difference in change in TG after 16 weeks of IP intake, in comparison to baseline
Difference in change in HDL-C after 16 weeks of IP intake, in comparison to baseline | 16 weeks
  Difference in change in HDL-C after 16 weeks of IP intake, in comparison to baseline
Difference in change in LDL-C after 16 weeks of IP intake, in comparison to baseline | 16 weeks
  Difference in change in LDL-C after 16 weeks of IP intake, in comparison to baseline
Difference in change in TC after 16 weeks of IP intake, in comparison to baseline | 16 weeks
  Difference in change in TC after 16 weeks of IP intake, in comparison to baseline
Difference in change in fasting blood glucose after 16 weeks of IP intake, in comparison to baseline | 16 weeks
  Difference in change in fasting blood glucose after 16 weeks of IP intake, in comparison to baseline
Difference in body fat mass (kg) change assessed per BIA after 4 weeks of IP intake, in comparison to baseline | 4 weeks
  Difference in body fat mass (kg) change assessed per BIA after 4 weeks of IP intake, in comparison to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Uebelhack, MD, Principal Investigator — Analyze & Realize
Locations (1):
- analyze & realize GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Uebelhack R, Bongartz U, Seibt S, Bothe G, Chong PW, De Costa P, Wszelaki N. Double-Blind, Randomized, Three-Armed, Placebo-Controlled, Clinical Investigation to Evaluate the Benefit and Tolerability of Two Dosages of IQP-AE-103 in Reducing Body Weight in Overweight and Moderately Obese Subjects. J Obes. 2019 Feb 3;2019:3412952. doi: 10.1155/2019/3412952. eCollection 2019. PMID 30863632